CLINICAL TRIAL: NCT01249781
Title: The Related Factors With Resilience in Caregivers Whose Child With Leukemia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: China Medical University Hospital (Other)
Responsible Party: China Medical University Hospital, China Medical University
Other Study IDs: DMR-99-IRB-191
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Condition 1. Children With ALL Are Still Alive and the Age of 18 Years of Age.; Condition 2. Has Been Completed to Guide the Treatment Regimen Were in Remission.; Condition 3. Caregiver Can or Taiwanese Language Communicator.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- resilience in caregivers whose child with ALL

SUMMARY:
The purpose of this study was to explore caregivers stress, family functioning, social support and family resilience of families whose children had acute lymphoblastic leukemia. The significantly correlation among caregivers stress, family functioning, social support and family resilience was also explored.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as acute lymphoblastic leukemia children, children with cancer are still alive and the age of 18 years of age.
2. Has been completed to guide the treatment regimen were in remission.
3. Caregiver can or Taiwanese language communicator.

Exclusion Criteria:

- Children with metastatic cancer who end chemical treatment of more than one year

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Families of children was diagnosed acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, No.2 Yuh Der Road, Taiwan